CLINICAL TRIAL: NCT05239429
Title: Improving the Mental Health & Well-Being of Healthcare Providers During the COVID-19 Pandemic: A Parallel Population Study Investigating the Reduction of Burnout and Enhancement of Well-Being Through the Transcendental Meditation Technique
Brief Title: Improving the Mental Health and Well Being of Healthcare Providers Through the Transcendental Meditation Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Clinical and Cosmetic Research (Other)
Collaborators: David Lynch Foundation (Other)
Responsible Party: Principal Investigator, Mark Steven Nestor, M.D., Ph.D., Director, The Center for Clinical and Cosmetic Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCCR 01-2020
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Burnout; Insomnia; Well Being
Keywords: Burnout; Well-being; Meditation; Insomnia
MeSH Terms: conditions — Burnout, Psychological; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcendental Meditation Technique (Experimental): Participants are trained on the use of the Transcendental Meditation Technique. They will perform the technique twice a day for 20-minutes per session.
  Interventions: Behavioral: Transcendental Meditation Technique
- Lifestyle-as-usual (control) (No Intervention): There is no change to the participants daily schedule and lifestyle.

INTERVENTIONS:
Behavioral: Transcendental Meditation Technique — Participants receive one-on-one training on how to use Transcendental Meditation technique which is then practiced twice daily for approximately 20 minutes.
  Arms: Transcendental Meditation Technique

SUMMARY:
The level of stress-related disorders experienced by Healthcare Providers (HCPs) has increased due to the recent COVID-19 Pandemic, impacting patient care and provider shortages. This trial aims to evaluate the use of the Transcendental Meditation Technique in improving burnout and wellbeing of HCPs over a 3-month trial period.

A total of 130 HCPs will be recruited from participating Miami hospitals, with 65 HCPs receiving training in the use of the Transcendental Meditation Technique. The remaining participants will be part of a matched control group and will not receive any training. Study outcomes will be assessed at baseline, 2 weeks, 1 month, and 3 months.

DETAILED DESCRIPTION:
This parallel population study aims to optimize and evaluate Healthcare Provider (HCP) wellness and performance through an evidence-based stress reduction program, Transcendental Meditation.

Transcendental Meditation (TM) has been found to be effective in reducing adverse mental health outcomes, including burnout, emotional exhaustion, depression, anxiety, insomnia, and trauma symptom severity. It is a mind-body program that allows the practitioner to experience progressively quieter, less excited states of mental activity.

For this trail, 65 HCPs affiliated with three participating Miami hospitals (Baptist Health South Florida Hospital, Mercy Miami Hospital and Encompass Health Rehabilitation Hospital of Miami) will receive instructions in the Transcendental Meditation Technique. A control group of similar numbers of HCPs will be recruited to match, to the best extent possible, for gender, age, type of HCP (doctor, nurse, etc.), and work schedule (e.g., days, nights, etc.). The control group participants will not receive Transcendental Meditation Technique training and will continue with their usual lifestyle.

The total duration of the study period will be 3 months. Study outcomes will be assessed at baseline, 2 weeks, 1 month, and 3 months' posttest, with change in burnout, insomnia, symptom, and well-being, as measured by the corresponding indexes as the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Fulltime healthcare providers, medical doctors, physician assistants, nurses or other HCPs involved in active patient care or administration of patient care (Hospital Administration).
2. 18 years or older.
3. Have treated COVID-19 patients or working at locations where COVID-19 patients are being treated.
4. Willing and able to complete both baseline and post-testing.
5. If being treated with psychoactive medications, the maintenance of a stable regimen for at least two months before enrollment.
6. In the non-control group, willing and able to dedicate the time to learning the Transcendental Meditation technique and practice it twice daily for approximately 20 minutes.

Exclusion Criteria:

1. Already instructed in the Transcendental Meditation technique.
2. Currently unstable psychiatric symptoms as demonstrated by self-report, medical chart, or psychiatric hospitalizations in the past six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Maslach Burnout Inventory- Human Services Survey (MBI-HSS) Score from Baseline | Baseline, 2 weeks, 1 month, and 3 months
  The Maslach Burnout Inventory- Human Services Survey (MBI-HSS) for Medical Personnel is used to measure participant burnout.
  The scale is a 22-item inventory with a seven-point response scale of 0-6 (0=never; 6= Every day).
Change from Baseline in Insomnia Severity Index (ISI) Score | Baseline, 2 weeks, 1 month, and 3 months
  The Insomnia Severity Index (ISI) scale contains 7 sleep-related questions to measure severity of sleep problems.
  A total score is calculated to interpret the participants level of insomnia, with a total score of 0-7 indicating no clinically significant insomnia and a score of 22-18 indicative of severe Clinical Insomnia.
Change from Baseline in Brief Symptom Inventory 18 (BSI 18) Score | Baseline, 2 weeks, 1 month, and 3 months
  The Brief Symptom Inventory 18 (BSI 18) is a 5-point rating scale used to gather patient-reported data to measure psychological distress and psychiatric disorders.
Change in Warwick-Edinburgh Mental Well Being Scale (WEMWBS) Score from Baseline | Baseline, 2 weeks, 1 month, and 3 months
  The Warwick-Edinburgh Mental Well Being Scale (WEMWBS) scale, covering both feeling and functioning aspects of mental wellbeing, contains 14 -items with 5 response categories, summed to provide a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nestor, M.D., Ph.D., Principal Investigator — Center for Clinical and Cosmetic Research
Locations (1):
- The Center for Clinical and Cosmetic Research, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: David Lynch Foundation Website — https://www.davidlynchfoundation.org/